CLINICAL TRIAL: NCT05200416
Title: A Randomized Cross-over Trial Investigating Heylo, a Novel App Driven Digital Supporting Ostomy Product
Brief Title: Investigation of Heylo, a Novel App Driven Digital Supporting Ostomy Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP345
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Ileostomy - Stoma; Colostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product - Heylo (Experimental): The arm includes the test product Heylo
  Interventions: Device: Heylo; Device: Standard of Care
- Standard of Care (Active Comparator): The arm includes Standard of Care
  Interventions: Device: Heylo; Device: Standard of Care

INTERVENTIONS:
Device: Heylo — Heylo is used in combination with the ostomy baseplate usually used by the subjects. It will detect and notify the subject of the occurrence of output leakage under an ostomy baseplate.
Device: Standard of Care — Standard of Care is the ostomy products (baseplate and bag) that the subject normally uses

SUMMARY:
People with intestinal stomas can have, despite development of better ostomy products, problems with leakage which influence their quality of life negatively.

To overcome this, Coloplast has developed a new supporting ostomy product called Heylo™, which has an adhesive sensor layer that should be placed underneath the baseplate. The sensor layer consists of an electronic sensor system that continuously detects moisture and output leakage underneath the baseplate. A transmitter connected to the sensor layer continuously evaluates the incoming information and sends a status to a smartphone software application, which based on a predefined flow decides which information to deliver to the user about the baseplate status.

The overall aim of this clinical investigation is to evaluate the benefits of the new supporting product, Heylo compared to Standard of Care.

DETAILED DESCRIPTION:
The Investigational device - Heylo, is already CE-marked.

The investigation is an open-labelled, randomized cross-over trial with two test periods evaluating Heylo and Standard of Care.

In total 144 subjects having an ileostomy or an colostomy will be included and randomized.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent to participate by signing the Informed Consent Signature Form.
* Is at least 18 years of age and has full legal capacity.
* Has an ileostomy or colostomy with consistent liquid/mushy fecal output (5-7 Bristol scale*)
* Is able to use one of the five test products (i.e. Ø40, Ø50, Ø60, Ø70, Ø80 mm).
* Has experienced leakage** under the baseplate at least three times within the last fourteen days. **Leakage defined as output seeping under the baseplate"
* Has worry about leakage to "some degree, high degree, or very high degree" (on a five-point Likert scale: Very low degree/Not at all, Low degree, some degree, High degree, very high degree)
* Is willing to refrain from use of ostomy paste.
* Has a smartphone compatible with the Heylo™ application
* Is able to follow study procedures for 4 months (assessed by investigator or delegate)

Exclusion Criteria:

* Is participating in other clinical investigations or has previously participated in this investigation
* Is pregnant or breastfeeding
* Has known hypersensitivity towards any of the products used in the investigation
* Is using/ has a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Ambe, Dr.med, Principal Investigator — GFO Kliniken Rhein Berg, Vinzenz Pallotti Hospital, 51429 Bergisch Gladbach-Bensberg, Germany
Locations (1):
- Peter C. Ambe, Bergisch Gladbach, Bergisch Gladbach,Nordrhein-Westfalen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ambe PC, Brunckhorst E, Hansen HD, Gotfredsen JL, Vestergaard M, Ajslev TA. Effect of a Novel Digital Leakage Notification System (Heylo) for Ostomy Care on Quality of Life and Burden of Living With an Intestinal Ostomy: The ASSISTER Trial, A Randomized Controlled Cross-Over Trial. Mayo Clin Proc Digit Health. 2023 Sep 1;1(3):438-449. doi: 10.1016/j.mcpdig.2023.06.013. eCollection 2023 Sep. PMID 40206623

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product - Heylo First, Then Standard of Care: Participants first used Heylo for 8 weeks ± 3 days. Then there was a cross-over and the participants used Standard of Care for 8 weeks ± 3 days.
  Heylo: Heylo is used in combination with the ostomy baseplate usually used by the subjects. It will detect and notify the subject of the occurrence of output leakage under an ostomy baseplate.
  Standard of Care: Standard of Care is the ostomy products (baseplate and bag) that the subject normally uses
  There was no 'Washout' period
- Standard of Care First, Then Test Product - Heylo: Participants first used Standard of Care for 8 weeks ± 3 days. Then there was a cross-over and the participants used Heylo for 8 weeks ± 3 days.
  Heylo: Heylo is used in combination with the ostomy baseplate usually used by the subjects. It will detect and notify the subject of the occurrence of output leakage under an ostomy baseplate.
  Standard of Care: Standard of Care is the ostomy products (baseplate and bag) that the subject normally uses
  There was no 'Washout' period
Period: First Intervention (8 Weeks ± 3 Days)
Arm/Group | Test Product - Heylo First, Then Standard of Care | Standard of Care First, Then Test Product - Heylo
Started | 72 | 72
Received Allocated Intervention | 71 | 72
Completed | 68 | 66
Not Completed | 4 | 6
Period: Second Intervention (8 Weeks ± 3 Days)
Arm/Group | Test Product - Heylo First, Then Standard of Care | Standard of Care First, Then Test Product - Heylo
Started | 68 | 66
Completed | 66 | 58
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Population: Due to the cross-over study design, all participants were randomized to receive all interventions. Baseline data has therefore been reported for all 'All Study Participants' (Intention-to-Treat Population).
  Intention-to-Treat Population included randomized participants who had been exposed to at least 1 product and with information on at least 1 endpoint (n=139).
  n=5 randomized participants only reported baseline data, and were not included in the ITT-Population.
Groups:
- All Study Participants: Due to the cross-over study design, all participants were randomized to receive all interventions. Baseline data has therefore been reported for all 'All Study Participants' being part of the Intention-to-Treat Population.
Arm/Group | All Study Participants
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 139

OUTCOME MEASURES:

1. Primary Outcome: Emotional Impact Score (Scale From 0-100)
Description: Measured by the validated OLI scale evaluated at the end of each test period. The questionnaire regarding Emotional impact contains 10 questions where the 4 answer options are: All of the time, Often, Sometimes and Rarely or never, which can be converted into a combined numerical score. The scale ranges from 0-100, where a score of 100 equals no impact and a score of 0 represents full impact.
Time Frame: 8 weeks
Population: The intention-to-treat (ITT) population (full analysis set) was constituted of all randomized subjects with valid informed consent who had been exposed to at least one product, and with information on at least one endpoint.
  Heylo --> Standard of Care: Analyzed (n=68) / Excluded from analysis (n=4) (Reasons: Only baseline data (n=4)).
  Standard of Care --> Heylo: Analyzed (n=71) / Excluded from analysis (n=1) (Reason: Only baseline data (n=1)).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Test Product - Heylo: The arm includes the test product Heylo
  Participants first used Heylo for 8 weeks ± 3 days. Then there was a cross-over and the participants used Standard of Care for 8 weeks ± 3 days.
  Heylo: Heylo is used in combination with the ostomy baseplate usually used by the subjects. It will detect and notify the subject of the occurrence of output leakage under an ostomy baseplate.
  Standard of Care: Standard of Care is the ostomy products (baseplate and bag) that the subject normally uses
- Standard of Care: The arm includes Standard of Care
  Participants first used Standard of Care for 8 weeks ± 3 days. Then there was a cross-over and the participants used Heylo for 8 weeks ± 3 days.
  Heylo: Heylo is used in combination with the ostomy baseplate usually used by the subjects. It will detect and notify the subject of the occurrence of output leakage under an ostomy baseplate.
  Standard of Care: Standard of Care is the ostomy products (baseplate and bag) that the subject normally uses
Arm/Group | Test Product - Heylo | Standard of Care
Number analyzed (Participants) | 139 | 139
score on a scale | 73.4 [68.9 to 77.9] | 62.0 [57.6 to 66.4]
Statistical Analysis 1: Comparison: Test Product - Heylo vs Standard of Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 11.42, 95% CI 2-sided [7.83 to 15.01]

2. Secondary Outcome: Participation in Society Domain Score (Scale From 0-100)
Description: Measured by WHODAS 2.0 evaluated at the end of each test period. The questionnaire regarding Participation in society contains 11 questions where the 5 answer options are: None, Mild, Moderate, Severe and Extreme or cannot do, which can be converted into a combined domain score. Each domain has a range of 0-100, where low scores equal better health and high scores indicate greater disability.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Test Product - Heylo | Standard of Care
Number analyzed (Participants) | 139 | 139
score on a scale | 33.0 [28.9 to 37.0] | 37.1 [33.1 to 41.2]
Statistical Analysis 1: Comparison: Test Product - Heylo vs Standard of Care; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.16, 95% CI 2-sided [-6.69 to -1.63]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the study period being 16 weeks ± 6 days.
Description: Mortality and Serious Adverse Events were assessed by investigators to not being related to the Test Product, nor Standard of Care.
Arm/Group | Test Product - Heylo | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/144 | 2/144
Serious Adverse Events (participants affected / at risk) | 3/144 | 4/144
Other Adverse Events (participants affected / at risk) | 5/144 | 0/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product - Heylo (N=144) | Standard of Care (N=144)
Morbus Crohn boost / new stoma (Surgical and medical procedures) | 0 | 1 — Product used: Standard of Care, Product: Not related, Procedure: Not related
Peritonitis (Surgical and medical procedures) | 0 | 1 — Product used: Standard of Care, Product: Not related, Procedure: Not related
Dysfunction of the gall bladder (Hepatobiliary disorders) | 1 | 0 — Product used: Heylo, Product: Not related, Procedure: Not related
Pneumonia (Infections and infestations) | 1 | 0 — Product used: Heylo, Product: Not related, Procedure: Not related
Prolapse (Surgical and medical procedures) | 0 | 1 — Product used: Standard of Care, Product: Not related, Procedure: Not related
Thyroid Surgery (Surgical and medical procedures) | 1 | 0 — Product used: Heylo, Product: Not related, Procedure: Not related
Early stoma re-operation (Surgical and medical procedures) | 1 | 0 — Product used: Heylo, Product: Not related, Procedure: Not related
Morbus Crohn boost (Surgical and medical procedures) | 0 | 1 — Product used: Standard of Care, Product: Not related, Procedure: Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product - Heylo (N=144) | Standard of Care (N=144)
Skin redness and irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 0 — Assessed by Investigator as having a causal relationship, or were probably or possibly related to Test Product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT05200416/Prot_SAP_000.pdf